CLINICAL TRIAL: NCT01926678
Title: Efficacy of Swedish Massage Therapy on Cancer-related Fatigue in Cancer
Brief Title: Efficacy of Swedish Massage Therapy on Cancer-related Fatigue in Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark H. Rapaport, Professor and Chairman, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00062853; R21AT007090 (NIH)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cancer Related Fatigue
Keywords: swedish massage; fatigue; light touch; inflammation
MeSH Terms: conditions — Fatigue; Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Swedish massage therapy (Experimental): Swedish massage therapy once per week for 6 weeks
  Interventions: Other: Swedish massage therapy
- Light touch therapy (Active Comparator): Light touch therapy once per week for 6 weeks
  Interventions: Other: Light touch therapy
- Wait list (Other): A 6 week wait list, followed by randomization to massage therapy or light touch therapy once per week for 6 weeks
  Interventions: Other: Swedish massage therapy; Other: Light touch therapy

INTERVENTIONS:
Other: Swedish massage therapy
  Arms: Swedish massage therapy; Wait list
Other: Light touch therapy
  Arms: Light touch therapy; Wait list

SUMMARY:
With approximately 12 million cancer survivors today in the United States alone, increased attention is being given to quality of life after cancer treatment. Cancer-related fatigue (CRF) is one of the most prevalent and debilitating symptoms experienced by people with cancer. It can persist for months or years after cancer therapy is completed and has a negative impact on all areas of function. Meaningful evidence-based treatment options for CRF are extremely limited and finding safe, inexpensive, and effective interventions for managing this distressing symptom are urgently needed. Basic research has shown that activation of the immune system can cause potent changes in behavior including reduced activity, fatigue, and decreased social behavior. Furthermore, research over the last decade has found a relationship between levels of CRF with increased inflammation. Thus, study of therapies that may decrease immune system activation in the setting of CRF represents a possible target for intervention. Massage therapy is one of the fastest growing alternative therapies and has a high rate of acceptance for symptom management among cancer patients. Massage has been shown in smaller studies with cancer patients to modulate the immune system. Moreover, massage has been demonstrated to significantly decrease markers of immune system activation in normal subjects. There are no published randomized controlled trials examining either the role of massage as an intervention primarily for CRF or investigating whether massage related decreases in immune system activation are responsible for improvement in CRF. This proposal investigates the effects of massage therapy on CRF among breast cancer survivors. The investigators' primary hypothesis is that Swedish Massage Therapy (SMT) will decrease CRF compared to a light touch condition and wait list control. The investigators' secondary hypothesis is that SMT will decrease CRF by reducing immune system activation. The investigators' main exploratory hypothesis is that a decrease in CRF will increase quality of life among cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women
* ages 18 to 65 (women above the age of 65 may be included at PI discretion)
* • with Stage 0-III breast cancer, status-post surgery treated with standard chemotherapy/chemoprevention and/or radiation.
* • Patients will be between 3 months and 4-years post treatment. Ongoing chemoprevention therapy is permissible. Based on ICD-10 proposed criteria, a diagnosis of CRF will require evidence from the history, physical exam, and laboratory findings that the fatigue is a consequence of cancer or cancer therapy and not primarily a consequence of comorbid psychiatric disorders (schizophrenia, depression, generalized anxiety disorder, bipolar disorder, dementia, delirium or OCD).
* Brief Fatigue Inventory (BFI) score of >25.
* Satisfactory results of screening safety labs, urine pregnancy test and drug test.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Women of reproductive capability will be enrolled, but each woman needs to discuss with the study team the method of birth control used and if the method is a reliable and effective method for her. If a woman becomes pregnant during the course of active study participation, she must agree prior to enrolling in the study that she will report the pregnancy to the study team. With a confirmed pregnancy, the subject will no longer receive the assigned treatment, but will continue to be followed per protocol.

Exclusion Criteria:

* Inability to lay supine for one hour at a time, given the nature of the massage intervention.
* Subjects who are actively suicidal or homicidal.
* Medical conditions felt to be clinically contributing to fatigue based on the investigator's history, physical examination, and assessment: anemia (hemoglobin less than 10 g/dl), hypothyroidism (thyroid stimulating hormone greater than 4.6 MCU/mL), uncontrolled pain, medical problems associated with fatigue: chronic obstructive pulmonary disease, congestive heart failure, renal disease, hepatic dysfunction, autoimmune disease, neurological disorders such as multiple sclerosis or Parkinson's disease, and sleep apnea.
* Medications felt to be clinically contributing to fatigue based on the investigator's history, physical examination, and assessment including: opioids, sedating anti-histamines, antidepressants, anxiolytics or neuroleptics.
* Body-mass index less than 18.5 (kg/m2).
* • Treatment with high dose systemic corticosteroids or continuous use of other immunosuppressants within the past 30 days.
* Unable to comply with the protocol for any reason.
* Use of non-steroidal anti-inflammatory drugs and aspirin is allowed but must be tracked.
* Other exclusion criteria include: illicit drug use, shift work, current dieting, excessive regular use of alcohol (more than two 5 ounce glasses of wine or equivalents/day) or a history of binge drinking (more than 7 drinks/24 hour period) within the last 6 months.
* Subjects who have used massage as a therapeutic modality (medical or psychological) at any point in their lives for the treatment of medical conditions.
* Subjects who have massages on a regular basis. Regular massage usage will be operationally defined as receiving 4 or more massages/year for the last 5 years.
* Subjects currently employing any other CAM manual therapy and/or holistic therapies to treat a perceived health problem. However, since past experience with CAM therapies should not confound any of the analyses of the experiments proposed in this study, we will not exclude individuals who have engaged in a CAM manual therapy in the past, nor will we exclude individuals who practice yoga or meditation for well-being, take vitamins or use nicotine.
* Adults over the age of 65 will generally be excluded from the study. This population tends to undergo changes in the physiological parameters we are evaluating. Therefore, inclusion of this population would skew various biological measures and this pilot investigation does not have a large enough sample size to control for such variability it. Older subjects could be included at the discretion of the PI.
* People unable to read and understand the informed consent document because of language difficulties.
* Women who are pregnant or lactating.
* Women who become pregnant while enrolled will be discontinued from the study and will be instructed to exercise, which is the standard recommendation for cancer-related fatigue. Inability or unwillingness of individual to give written informed consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cancer-Related Fatigue | 6 weeks
  The primary aim of this study is to determine whether a 6-week Swedish massage therapy (SMT) intervention can decrease cancer-related fatigue, as measured by the Multidimensional Fatigue Inventory (MFI), among breast cancer survivors who have received both radiation and chemotherapy and have CRF. We hypothesize that SMT will decrease fatigue more than light touch (LT) or a wait list control (WLC) condition as assessed by the MFI.

SECONDARY OUTCOMES:
Inflammation | 6 weeks
  A secondary aim of this study is to determine whether the hypothesized decrease in cancer-related fatigue is due to Swedish massage therapy modulating the immune system of subjects with cancer-related fatigue to decrease chronic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Rapaport, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States